CLINICAL TRIAL: NCT01375816
Title: A Randomized Phase II Study of PEP02 or Irinotecan in Combination With Leucovorin and 5-Fluorouracil in Second Line Therapy of Metastatic Colorectal Cancer
Brief Title: Liposome-encapsulated Irinotecan Hydrochloride PEP02 or Irinotecan Hydrochloride, Leucovorin Calcium, and Fluorouracil as Second-Line Therapy in Treating Patients With Metastatic Colorectal Cancer
Acronym: PEPCOL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: efficacy interim analysis as per protocol
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000701454; FRE-GERCOR-PEPCOL-C10-1; EU-21115; EUDRACT-2010-020468-39; PHARMAENGINE-FRE-GERCOR-PEPCOL
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFIRI 1 or m FOLFIRI3-Bevacizumab (Active Comparator): FOLFIRI 1-Bevacizumab:
  Day 1 H0 : Bevacizumab 5 mg/kg, 30-90 min infusion H+1: Irinotecan 180 mg/m² in 250 ml NaCl 0.9%, 1h infusion Folinic Acid 400 mg/m² (l + d racemic form, or l form 200 mg/m²) over 2h H + 3: 5-FU bolus 400 mg/m², 15 min infusion H + 3.5: 5-FU continuous infusion 2400 mg/m² 46-h infusion End of cycle: day 14
  modified FOLFIRI3-Bevacizumab H0 :Bevacizumab 5 mg/kg, 30-90 min infusion H+1:Irinotecan 90 mg/m² in 250 ml NaCl 0.9%, 1h infusion H+1: Folinic Acid 400 mg/m² (l + d racemic form, or l form 200 mg/m²) 2-h infusion H + 3: 5-FU continuous infusion 2400 mg/m² 46-h infusion Day 3 (H+49) H0 Irinotecan 90 mg/m² in 250 ml NaCl 0.9%, 1h infusion End of cycle: day 14
  Interventions: Drug: FOLFIRI 1-Bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: Bevacizumab
- FUPEP-Bevacizumab (Experimental): Day 1 H0 :Bevacizumab 5 mg/kg, 30-90 min infusion H +1 :PEP02 80 mg/m² , 1h30 infusion. The infusion time could be reduced to 1h from cycle 2 if no acute infusion reaction has occured in cycle 1.
  H +1 : Folinic Acid 400 mg/m² (l + d racemic form, or l form 200 mg/m²) , 2-h infusion H +3 : 5-FU continuous infusion 2400 mg/m² 46-h infusion End of cycle: day 14
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: liposome-encapsulated irinotecan hydrochloride PEP02; Drug: Bevacizumab

INTERVENTIONS:
Drug: FOLFIRI 1-Bevacizumab
  Arms: FOLFIRI 1 or m FOLFIRI3-Bevacizumab
Drug: fluorouracil
Drug: irinotecan hydrochloride
  Arms: FOLFIRI 1 or m FOLFIRI3-Bevacizumab
Drug: leucovorin calcium
Drug: liposome-encapsulated irinotecan hydrochloride PEP02
  Arms: FUPEP-Bevacizumab
Drug: Bevacizumab

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposome-encapsulated irinotecan hydrochloride PEP02, irinotecan hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving liposome-encapsulated irinotecan hydrochloride PEP02 together with leucovorin calcium and fluorouracil is more effective than giving irinotecan hydrochloride together with leucovorin calcium and fluorouracil as second-line therapy in treating patients with metastatic colorectal cancer.

PURPOSE: This randomized phase II trial is studying liposome-encapsulated irinotecan hydrochloride PEP02 given together with leucovorin calcium and fluorouracil to see how well it works compared with giving irinotecan hydrochloride together with leucovorin calcium and fluorouracil as second-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the objective response rates (complete response and partial response) in patients with metastatic colorectal cancer treated with liposome-encapsulated irinotecan hydrochloride PEP02, leucovorin calcium, and fluorouracil (FUPEP) Versus irinotecan hydrochloride, leucovorin calcium, and fluorouracil (FOLFIRI 1) or leucovorin calcium, fluorouracil, and irinotecan hydrochloride-modified (FOLFIRI 3-modified).

Secondary

* To determine the safety of these regimens in these patients.
* To determine progression-free survival of these patients.
* To determine overall survival of these patients.
* To assess the quality of life of these patients.
* To assess the correlation of UGT1A family polymorphism and the toxicity of liposome-encapsulated irinotecan hydrochloride PEP02 or irinotecan hydrochloride.

OUTLINE: This is a multicenter study. Patients are stratified, in terms of prognosis, according to treatment center, prognostic score (ECOG performance status [PS] 0 and normal LDH value vs ECOG PS > 1 and/or LDH > 1 times upper limit of normal), and time to progression after first-line therapy (≥ 9 months vs < 9 months). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are assigned to either the FOLFIRI 1 or Modified FOLFIRI 3 treatment groups according to the investigator's discretion in combination with bevacizumab

  * FOLFIRI 1 in combination with bevacizumab: Patients receive bevacizumab over 30-90 minutes,irinotecan hydrochloride over 1 hour and leucovorin calcium IV over 2 hours on day 1 and a bolus of fluorouracil followed by fluorouracil IV over 46 hours beginning on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity
  * Modified FOLFIRI 3 in combination with bevacizumab: Patients receive bevacizumab,irinotecan hydrochloride, leucovorin calcium, and fluorouracil as in FOLFIRI 1. Patients also receive irinotecan hydrochloride IV over 1 hour on day 3. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
* Arm II (FUPEP)in combination with bevacizumab: Patients receive bevacizumab over 30-90 minutes liposome-encapsulated irinotecan hydrochloride PEP02 IV over 60-90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacogenetic analysis of UGT1A family polymorphisms. Quality of life is assessed by using a generic scale EQ-5D and the QLQ-C30 questionnaire at baseline and after courses 4 and 8.

After completion of study treatment, patients are followed up at day 30 and then every 2-3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS

* Histologically proven adenocarcinoma of colon or rectum

  * Metastatic disease, exclusive of bone metastasis
  * Not suitable for complete carcinological surgical resection
* Patients regardless KRAS status (wild type or mutated) or previous anti EGFR treatment or not.
* Measurable lesion (greater than 1 cm) as assessed by CT scan or MRI according to RECIST criteria (version 1.1)
* Must have received prior oxaliplatin-based chemotherapy for metastatic disease
* No symptomatic ascites or pleural effusion not evacuated prior to study entry
* No history or evidence of CNS metastasis

PATIENT CHARACTERISTICS:

* WHO or ECOG performance status 0-2
* Absolute neutrophil count greater than 1500 per mm3
* Platelet count greater than 100 000 per microL
* Hemoglobin greater than 9 g per dL (may be transfused to maintain or exceed this level)
* INR less or equal than 1.5. aPTT less than 1.5 ULN (exemption:patients on full anticoagulation due to VTE must have an in-range INR.
* Serum creatinine less than 150 micromol per L
* Calculated creatinine clearance greater than 30 mL per min
* Total bilirubin less than 1.5 times upper limit of normal
* Proteinuria less than 2 plus (dipstick urinalysis) or less than 1 g per 24 hours.
* Negative serum pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe arterial thromboembolic events within the past 6 months, including myocardial infarction and stroke
* No baseline diarrhea greater than grade 1
* No total or partial bowel obstruction
* No uncontrolled hypercalcemia
* No uncontrolled hypertension, or history of hypertensive crisis, or hypertensive encephalopathy
* No other prior or concurrent malignancy, except adequately treated in situ carcinoma of the uterine cervix, basal cell or squamous cell carcinoma of the skin, or cancer in complete remission for more than 5 years
* No other serious and uncontrolled non-malignant disease
* Major surgery or traumatic injury within the last 28 days.
* No known allergy to any excipients of study drugs
* Must be registered in a national health care system (CMU included)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior anti-EGFR therapy allowed
* No prior irinotecan hydrochloride
* No concurrent agents known to have anticancer activity
* No concurrent radiotherapy
* No participation in another clinical trial with any investigational drug or treatments concurrently or within the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Tumor response | at 2 months
  Assessment of tumor response at 2 month after randomization by RECIST 1.1

SECONDARY OUTCOMES:
Safety | before each 2-weeks cycles
  assessment of adverse events and toxicity according NCI CTC v4.0
Progression-free survival | the time from the date of randomization to the date of progressive disease (RECIST criteria) or death (any cause)
Overall survival | from the date of randomization to the date of patient death, due to any cause, or to the last date the patient was known to be alive
Quality of life | at baseline, cycle 4, and cycle 8
  Quality of life will be assessed by using a generic scale EQ-5D and the QLQ-C30 questionnaire
Correlation of UGT1A family polymorphism and the toxicity of liposome-encapsulated irinotecan hydrochloride PEP02 or irinotecan hydrochloride | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Maindrault-Goebel, MD, Principal Investigator — Hopital Saint Antoine
Locations (1):
- Hopital Saint Antoine, Paris, France